CLINICAL TRIAL: NCT01246128
Title: PET Assay of Acetylcholine Beta2* Nicotinic Receptor Density in Smoking and Non-Smoking Schizophrenics
Brief Title: Nicotinic Receptor Density in Smoking and Nonsmoking Schizophrenics
Status: Withdrawn | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999911463; 11-DA-N463
Record Dates: First submitted 2010-11-20; First posted 2010-11-23 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-07-12

CONDITIONS: Schizophrenia
Keywords: Nicotinic Acetylcholine Receptors; Schizophrenia Smokers; PET Imaging
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
Background:

- Previous studies have suggested that smoking cigarettes affects the number of receptors in the brain for nicotine, a chemical present in cigarette smoke. The receptors play a role in an individual's ability to think and concentrate. Many people with schizophrenia and similar disorders smoke, and research suggests that smoking may temporarily improve concentration and focus in individuals with schizophrenia. Researchers are interested in studying both current smokers and nonsmokers with schizophrenia to determine whether smoking affects the number of nicotine receptors in the brains of people with schizophrenia.

Objectives:

- To study the distribution and volume of nicotine receptors in the brains of individuals with schizophrenia who are either nonsmokers or current smokers.

Eligibility:

* Individuals between 18 and 50 years of age who have been diagnosed with schizophrenia and are either nonsmokers or current smokers (at least 10 cigarettes per day for the past year).
* Current smokers must be able to give up smoking for 48 hours.

Design:

* This study involves an initial screening visit and up to five study visits.
* After the screening visit, participants will have two sessions in which they will complete questionnaires about thoughts, memory, and smoking habits. Smokers will also have nicotine blood and carbon monoxide breath levels taken during these sessions, before and after smoking a cigarette.
* Participants will have sessions with imaging studies (e.g., magnetic resonance imaging) to provide baseline measurements for later tests, and will also have tests to measure brain electrical activity.
* Participants will have a positron emission tomography (PET) scanning session to examine the nicotine receptors in the brain. Participants will need to stay overnight (nonsmokers) or for 2 nights (smokers) as an inpatient before the session. The PET scan session will take up to 6 hours, although participants will only be in the scanner for up to 3 hours.
* Participants will have a follow-up phone call with study researchers 1 week after the PET scanning session.

DETAILED DESCRIPTION:
Objective:

The objective of this study is to determine the distribution and volume of distribution (Vt) in vivo of Beta2* acetylcholine receptors (Beta2* nAChR) in schizophrenic smokers and nonsmokers and compare this to published data from normal healthy subjects who are smokers and nonsmokers.

Study population:

Participants will be volunteers with a diagnosis of schizophrenia aged 18 to 50 years. The proposed sample size is 10 per group: nonsmokers or ex-smokers and smokers for a total of 20 participants.

Design:

One PET study lasting up to 8 hours after combination of bolus and continuous infusion administration of 2[(18)F] FA-85380. Smokers will be abstinent for at least 48 hrs. Subjects will also undergo a structural MRI scan for purposes of registration of PET scan data.

Outcome Measures:

Data from 20 schizophrenic patients (10 smokers and 10 nonsmokers) will be compared to published data from healthy controls. Total volume of distribution (VT) which is a measure of receptor density and distribution of Beta2 nAChR* will be determined in Schizophrenic smokers and nonsmokers and differences in these values will be compared to published values for the differences in nicotinic acetylcholine receptor density in healthy smokers and nonsmokers (Mukhin et al., 2008) Also, receptor distribution and VT will be correlated with levels of smoking and symptom profiles in the schizophrenic patients studied.

ELIGIBILITY:
* INCLUSION CRITERIA:

Age: Subjects will be male and female volunteers aged 18 to 50 years.

Contact: All subjects must have a stable point of contact and must agree to participate in one PET study and one MRI scan.

Smoking group: must smoke at least 10 cigarettes per day for at least the last year. They should have experience with abstaining from smoking for at least 48 h.

Nonsmoking group: Subjects in the non-smoking group must be nonsmokers or have smoked less than 100 cigarettes in their lifetime and have ceased smoking at least two years before the start of the study.

Diagnosis: Each volunteer will have a diagnosis of schizophrenia using DSMIV criteria. Each subject will have the following information available for diagnostic consideration: Structured Clinical Interview for DSM-IV Axis I Disorders (SCID-I), a general psychiatric interview for past illness characteristics and family history, information from 2-3 months of independent clinician observation including current detailed mental status evaluations using the Brief Psychiatric Rating Scale (BPRS), Schedule for the Assessment of Positive and Negative Symptoms (SAPS/SANS), and Schedule for Deficit Syndrome (SDS). An assessment of impulsivity will also be done (Patton, 1995).

Comorbidity: No subject with a current axis I diagnosis other than schizophrenia will be allowed. No subject with known claustrophobia will be allowed.

Medications: Study participants will continue to take their antipsychotic medications that they have been taking for at least 3 months prior to the study. Haldol, risperidone and olanzapine will be allowed because of their lack of significant effect on the density of beta2* nACh receptors after prolonged administration to rats (Haldol; Breese et al., 2000; risperidone and olanzapine; personal communication, Mukhin, also SFN abstract).

EXCLUSION CRITERIA:

Weight: Anyone weighing more than 300 lbs is excluded from the study. The purpose of this exclusion is the weight limit of the PET scanner.

History of Drug Abuse: Participants reporting current or having a significant history of illicit drug abuse will be excluded from the study. Subjects may use moderate amounts of alcohol and caffeine and smoke an occasional marijuana cigarette, but must not be dependent on alcohol, caffeine or marijuana. No alcohol or marijuana for at least 72 hours prior to scanning. No smoking for 48 hrs before the PET scan.

Current Medication Use: Participants will continue to use their prescription medications. The following hypertension medications will be exclusionary: Indapamide, spironolactone, clonidine, guanfacine, methyldopa, propranolol. Over the counter medications are not exclusionary, however, subjects will not be allowed to use over the counter medications in the week prior to their PET scan.

CNS disease: History of known structural brain abnormalities (e.g., neoplasm, subarachnoid cysts), cerebrovascular disease, infectious disease (e.g., abscess), history of head trauma (defined as documented loss of consciousness for 5 min or greater), history of seizures as an adult, sleep apnea.

Cardiovascular, pulmonary, or systemic disease: Untreated hypertension known arrhythmia, symptomatic or known coronary artery disease; history of endocarditis, cerebral embolism, obstructive pulmonary disease, asthma, active tuberculosis, known endocrine disease (derangements in adrenal, thyroid, bone or reproductive function) known chronic renal or hepatic dysfunction, known HIV seropositive, known current autoimmune disease involving the CNS, type I diabetes mellitus. Subjects with type II diabetes mellitus will be allowed if their Hb A1C is less than 7.

Special considerations for female subjects. Female participants who are planning to become pregnant, currently pregnant or nursing will not be allowed to participate in this study because of potential damage to the fetus or baby from the radiation. In addition, women of child bearing age who are sexually active are required to use an effective form of birth control for the duration of the study. Effective forms of birth control include:

1. hormonal contraceptives (birth control pills, injectable hormones, vaginal ring hormones),
2. surgical sterility (tubal ligation or hysterectomy)
3. IUD
4. Diaphragm with spermicide
5. Condom with spermicide

Female subjects will be given a serum pregnancy test (quantitative beta HCG) within 24 hours of the PET study. Menstrual cycle phase or sex has not been shown to affect receptor availability (Cosgrove et al., 2007).

Radiation exposure: Any subject who has participated in any research studies in which he/she received a radiation exposure that would result in combination with the present study, in a total effective radiation exposure (from research studies) exceeding 5.0 rem in a year.

Children under the age of 18 will be excluded to avoid unnecessary exposure to radiation to these populations.

Presence in body of metallic implants or materials that could be moved by the magnet of the MRI scanner: pacemakers, surgical implants, aneurysm clips, dental braces, bullet(s) or other metallic materials.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2010-10-31; Study Completion 2011-07-12

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Johns Hopkins University, Baltimore, Maryland
  - Maryland Psychiatric Research Center (MPRC) 55 Wade Avenue, Catonsville, Maryland

REFERENCES:
- [Background] Adler LE, Hoffer LJ, Griffith J, Waldo MC, Freedman R. Normalization by nicotine of deficient auditory sensory gating in the relatives of schizophrenics. Biol Psychiatry. 1992 Oct 1;32(7):607-16. doi: 10.1016/0006-3223(92)90073-9. PMID 1450287
- [Background] Adler LE, Hoffer LD, Wiser A, Freedman R. Normalization of auditory physiology by cigarette smoking in schizophrenic patients. Am J Psychiatry. 1993 Dec;150(12):1856-61. doi: 10.1176/ajp.150.12.1856. PMID 8238642
- [Background] Bottlaender M, Valette H, Roumenov D, Dolle F, Coulon C, Ottaviani M, Hinnen F, Ricard M. Biodistribution and radiation dosimetry of 18F-fluoro-A-85380 in healthy volunteers. J Nucl Med. 2003 Apr;44(4):596-601. PMID 12679405